CLINICAL TRIAL: NCT02158052
Title: Combined HLA-Matched Bone Marrow and Kidney Transplantation for Multiple Myeloma or Other Hematologic Disorders With End Stage Renal Disease
Brief Title: Combined Bone Marrow and Renal Transplantation for Hematologic Disorders With End Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas Spitzer, Director, Bone Marrow Transplant Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KdBMT-2
Record Dates: First submitted 2014-05-30; First posted 2014-06-06 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma; Amyloidosis
Keywords: HLA matched; bone marrow transplantation; kidney transplantation
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis | interventions — Tacrolimus; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone Marrow and Kidney RECIPIENTS (Experimental): combined bone marrow and kidney transplantation
  Interventions: Drug: Tacrolimus; Drug: Equine Anti-thymocyte globulin; Procedure: Kidney transplant from a related donor; Drug: Bone marrow transplant from a related donor; Radiation: Total body irradiation 400 centigray (200 cGy X 2)
- Bone Marrow and Kidney DONORS (Other): Donors who donate bone marrow and kidney
  Interventions: Procedure: Kidney transplant from a related donor

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus starting on Day -1
  Arms: Bone Marrow and Kidney RECIPIENTS
Drug: Equine Anti-thymocyte globulin — 20 mg/kg IV on Days -3, -1, +1, +3
  Arms: Bone Marrow and Kidney RECIPIENTS
Procedure: Kidney transplant from a related donor — On Day 0 the renal transplant is performed according to standard surgical techniques.
Drug: Bone marrow transplant from a related donor — Donor bone marrow (> 2 x 10e8 nucleated cells/kg of recipient body weight) is prepared for infusion according to the standard procedure. The infusion begins in the operating room as soon as the vascular anastomosis of the renal allograft has been completed.
  Arms: Bone Marrow and Kidney RECIPIENTS
Radiation: Total body irradiation 400 centigray (200 cGy X 2) — On transplant day -1
  Arms: Bone Marrow and Kidney RECIPIENTS

SUMMARY:
This pilot trial offers the unique opportunity for both the treatment of multiple myeloma or systemic AL amyloidosis for which hematopoietic stem cell transplantation would be ordinarily indicated and the reversal of end-stage renal failure, while avoiding the risks associated with long-term standard anti-rejection therapy used in renal transplantation. The primary objectives of this study are to assess renal allograft tolerance (that is, the acceptance of the kidney without the need for anti-rejection therapy), assess anti-tumor response rates in multiple myeloma and AL amyloidosis, and assess complication rates for genetically (HLA) matched related donor combined bone marrow and kidney transplantation using a low dose total body irradiation based preparative regimen.

DETAILED DESCRIPTION:
The induction of transplantation tolerance involves the specific elimination of the immune response to the transplant but not to other antigens. In the realm of kidney transplantation, tolerance means that the recipient is unable to detect the donor transplant kidney as foreign, and therefore the recipient is unable to reject the kidney. Donor bone marrow engraftment leads to kidney graft tolerance in animal models. Renal failure is a major complication of multiple myeloma and AL amyloidosis for which the only known cure is allogeneic bone marrow transplantation. Standard bone marrow transplantation is associated with prohibitive toxicities in patients with end stage renal disease, and is generally not considered an option for those patients. Patients with multiple myeloma and AL amyloidosis are excluded from conventional renal transplantation protocols because of their underlying malignancy. A less toxic bone marrow transplantation protocol, utilizing low dose total body irradiation and anti-thymocyte globulin, combined with renal transplantation, could provide an opportunity for cure of the myeloma or amyloidosis and correction of end stage renal disease. In addition, successful marrow engraftment may be expected to lead to a state of tolerance. Successful implementation of tolerance would be a major benefit to transplant recipients. The significance of developing tolerance is that the patient could be spared the disabling complications of indefinite immunosuppression, which include infections, cataracts, osteoporosis, diabetes, atherosclerosis, hypertension, and malignancy.

ELIGIBILITY:
Participant Inclusion Criteria

* Participants with end-stage renal failure due to or in association with multiple myeloma or systemic AL amyloidosis which hematopoietic cell transplantation is appropriate and a ≥ 50% five-year survival probability with transplantation is expected. This includes, but is not limited to:
* Multiple myeloma (MM), ISS stage II or III in complete or very good partial remission
* AL amyloidosis without significant cardiac disease
* Males or females 18 - 65 years of age.
* Participants must have an HLA-matched or one of six HLA A, B, or DR antigen-mismatched related donor, with high resolution molecular class I and II allele typing.
* Men and women of reproductive potential must agree to use a reliable method of birth control during the treatment, and women should do so for a period of 2 years following the transplant.
* Participants should be on dialysis or have a CrCl <20 ml/min.
* Patients should not have evidence of renal recovery of their renal failure over a 90 day period of therapy for their underlying malignancy or other blood disorder.
* .
* Patients with a history of other malignancies excluding basal cell carcinoma of the skin and carcinoma in situ of the cervix with a disease-free survival interval of >2 years. Patients with the following malignancies must demonstrate a 5 year disease-free survival:

  * Breast cancer with positive nodes
  * Malignant melanoma (other than in situ)
  * Colorectal cancer (other than Dukes Stage A or B1)
* Patients with multiple myeloma must have received previous treatment with a bortezomib-based regimen.

Patients with AL amyloidosis must have received previous treatment with a bortezomib-based regimen and/or autologous stem cell transplantation

* Patients with a history of malignant melanoma must be reviewed by an independent oncologist prior to enrollment.
* Recipient ability to understand and provide informed consent.

Participant Exclusion Criteria

* Evidence of active infection as defined by: a) clinical syndrome consistent with viral or bacterial infection (e.g., influenza, URI, UTI) or b) fever with a clinical site of infection identified, or c) microbiologically documented infection, including, but not limited to, bacteremia or septicemia.
* Participation in other investigational drug use at the time of enrollment.
* Contraindication to therapy with any one of the proposed agents (e.g., history of allergy to horse serum in ATG).
* Serologic positivity to HIV or HCV.
* Women of childbearing age in whom adequate contraception cannot be maintained.
* AST/ALT > 3 x normal or bilirubin > 1.5 x normal (unless due to Gilbert's syndrome).
* Pregnancy or uncontrolled serious medical illness not related to underlying myeloma.
* Cardiac ejection fraction < 40% by echocardiogram.
* FEV1 < 50% predicted or corrected DLCO < 50% predicted.
* ABO blood group incompatibility in the host-vs-graft direction.

  * Diagnosis of myelodysplastic syndrome

Donor Inclusion Criteria

* HLA-matched or one of six HLA A, B, or DR antigen-mismatched related male or female donor 18-65 years of age.
* ECOG performance status 0 or 1.
* Excellent health per conventional pre-donor history (medical and psychosocial evaluation).
* Acceptable laboratory parameters (hematology in normal or near-normal range; liver function < 2 times the upper limit of normal and normal creatinine).
* Compatible ABO blood group.
* Negative donor lymphocyte crossmatch.
* No positive testing for viral infection (HbsAg, HIV, HCV, HTLV-1).
* Cardiac/Pulmonary evaluation within normal limits (CXR, EKG).
* Donor ability to understand and provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-02; Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Spitzer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD, including the study protocol and consent form with other researchers.
  Any publication that results from this trial will not include any patient identifiers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow and Kidney RECIPIENTS: Single arm combined bone marrow and kidney transplantation
  Tacrolimus: Tacrolimus starting on Day -1
  Equine Anti-thymocyte globulin: 20 mg/kg IV on Days -3, -1, +1, +3
  Kidney transplant from a related donor: On Day 0 the renal transplant is performed according to standard surgical techniques.
  Bone marrow transplant from a related donor: Donor bone marrow (> 2 x 10e8 nucleated cells/kg of recipient body weight) is prepared for infusion according to the standard procedure. The infusion begins in the operating room as soon as the vascular anastomosis of the renal allograft has been completed.
  Total body irradiation 400 centigray (200 cGy X 2): On transplant day -1
- Bone Marrow and Kidney DONORS: Donor nephrectomy and bone marrow harvest (> 2X10e8/kg nucleated cells/kg recipient body weight) on Day 0
Period: Overall Study
Arm/Group | Bone Marrow and Kidney RECIPIENTS | Bone Marrow and Kidney DONORS
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 transplant recipient and their donor were enrolled.
Groups:
- Bone Marrow and Kidney RECIPIENT: Single arm combined bone marrow and kidney transplantation
  Tacrolimus: Tacrolimus starting on Day -1
  Equine Anti-thymocyte globulin: 20 mg/kg IV on Days -3, -1, +1, +3
  Kidney transplant from a related donor: On Day 0 the renal transplant is performed according to standard surgical techniques.
  Bone marrow transplant from a related donor: Donor bone marrow (> 2 x 10e8 nucleated cells/kg of recipient body weight) is prepared for infusion according to the standard procedure. The infusion begins in the operating room as soon as the vascular anastomosis of the renal allograft has been completed.
  Total body irradiation 400 centigray (200 cGy X 2): On transplant day -1
- Bone Marrow and Kidney DONOR: Kidney transplant from a related donor: On Day 0 the renal transplant is performed according to standard surgical techniques.
  Bone marrow transplant from a related donor: Donor bone marrow (> 2 x 10e8 nucleated cells/kg of recipient body weight) is prepared for infusion according to the standard procedure.
- Total: Total of all reporting groups
Arm/Group | Bone Marrow and Kidney RECIPIENT | Bone Marrow and Kidney DONOR | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53 [53 to 53] | 46 [46 to 46] | 49.5 [46 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Renal Allograft Rejection at 6 Months Post-transplant
Description: The Primary Outcome is: the incidence of renal allograft rejection at 6 months post-transplant
Time Frame: 6 Months
Population: One bone marrow/kidney transplant recipient was enrolled and treated on this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow and Kidney RECIPIENTS
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Anti-Tumor Response Rate
Description: This is measurement is summarized via bone marrow biopsy results and blood assays through 3 years.
  Anti-tumor response is assessed according to Center for International Blood and Marrow Transplant Research (CIBMTR.org) criteria.
  For multiple myeloma, based on assessment of serum and urine immunofixation, the presence or absence of soft tissue plasmacytomas and analyses of bone marrow aspirate and biopsy samples, response categories include stringent complete remission (sCR), complete remission (CR), near CR (nCR) very good partial response (VGPR), partial response (PR), stable disease (SD), and progressive disease (PD).
  For AL amyloidosis, based on assessment of serum and urine immunofixation and serum free light chain ratio, hematologic response categories include complete response, very good partial response, partial response, no response/stable disease and progressive disease. Organ responses are also assessed according to organ specific criteria.
Time Frame: 3 years
Population: One bone marrow/kidney recipient was enrolled and treated on this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow and Kidney RECIPIENTS
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 years
Description: Adverse event information was assessed by study investigators and entered into an internal Bone Marrow Transplant database.
Arm/Group | Bone Marrow and Kidney RECIPIENT | Bone Marrow and Kidney DONOR
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow and Kidney RECIPIENT (N=1) | Bone Marrow and Kidney DONOR (N=1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA — Transient acute kidney injury due to tacrolimus and engraftment syndrome
Hematopoietic graft rejection (Blood and lymphatic system disorders) | 1 (1) | NA — Delayed (secondary) hematopoietic graft rejection. A second HLA-matched related stem cell transplant was performed from the same donor on 5/11/16 with successful and sustained engraftment.
Aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Pulmonary aspergillosis following hematopoietic graft rejection, treated to resolution following a second hematopoietic cell transplant from the same donor and anti-fungal therapy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow and Kidney RECIPIENT (N=1) | Bone Marrow and Kidney DONOR (N=1)
Perinephric hematoma (Renal and urinary disorders) | 1 (1) | NA — A postoperative transient perinephric hematoma occurred, not requiring surgical intervention.
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA — Abdominal pain due to constipation occurred which was alleviated by a bowel regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02158052/Prot_SAP_000.pdf